CLINICAL TRIAL: NCT06901310
Title: Effectiveness of Recruitment, Retention Strategies, and Data Collection Quality: A Feasibility Study in Combat Athletes With Mild Traumatic Brain Injury
Brief Title: A Feasibility Study in Combat Athletes With Mild Traumatic Brain Injury
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Harl (Other)
Responsible Party: Sponsor-Investigator, Michael Harl, Physician - Plastic Surgery, Marshfield Clinic Research Foundation
Organization: Marshfield Clinic Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAR10123
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-05

CONDITIONS: Mild Traumatic Brain Injury (mTBI); Brain Injury; Concussion
Keywords: brain injury; concussion; Mild traumatic brain injury (mTBI)
MeSH Terms: conditions — Brain Concussion; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HBOT Treatment Group (Experimental)
  Interventions: Device: Hyberbaric Oxygen Therapy
- Conventional Rest Control Group (No Intervention)

INTERVENTIONS:
Device: Hyberbaric Oxygen Therapy — Treating participants with 100% Oxygen at 2.4 Atmospheres for 90 minutes at 10 treatments.
  Arms: HBOT Treatment Group

SUMMARY:
The use of Hyberbaric Oxygen Therapy (HBOT) would be a new treatment plan rather than conventional rest. If effective, this new use technology would add to the clinical treatment among mild traumatic brain injury (mTBI) patients. The use of a point of care Glial Fibrillary Acidic Protein (GFAP) biomarker would aid in clinical decision making to create a new care plan of return to sport among unarmed combat athletes who suffer from mTBI. The innovation would be a new treatment and diagnosis strategy that will protect these athletes from serious long-term sequelae. There are no published randomized controlled studies using HBOT to treat concussed athletes within one week of injury. There are no published studies using GFAP levels to predict post concussive symptoms (PCS).

ELIGIBILITY:
Inclusion Criteria:

* 18 Years or older
* Male Unarmed Combat Athlete
* 30-day suspension (head injury without technical knockout or incapacitation)
* 60-day suspension (head injury with technical knockout or incapacitation)
* 90-day suspension (head injury with loss of consciousness)

Exclusion Criteria:

* Prisoner status
* Female
* Suspension group injury severity would not include moderate to severe GCS <13

These suspension groups are not based on GCS; therefore, GCS is not part of the inclusion criteria. This group will be divided into randomized groups, patients who will be treated with HBOT and patients who will receive the standard of care, which is rest.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact Neurological Scores | 13 Weeks
  The Impact scores are a percentile 1% to 100%. Any score under 50% is considered a need for neurological or primary care consultation for a concussion

CONTACTS AND LOCATIONS:
Locations (1):
- Marshfield Clinic, Marshfield, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No